CLINICAL TRIAL: NCT02683707
Title: The Platelet Aggregation After tiCagrelor Inhibition and FentanYl Trial
Brief Title: The Platelet Aggregation After tiCagrelor Inhibition and FentanYl Trial (PACIFY)
Acronym: PACIFY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00089755
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Blood Platelets; Fentanyl
MeSH Terms: conditions — Coronary Artery Disease | interventions — Fentanyl; Lidocaine; Midazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCI without IV opiate (Experimental): IV midazolam and Local Anesthetic, with removal of IV fentanyl from peri-procedural analgesia (which is otherwise routinely given)
  Interventions: Other: Removal of Fentanyl from peri-procedural analgesia; Drug: Lidocaine; Drug: Midazolam
- PCI with IV opiate (Active Comparator): IV midazolam and Local Anesthetic and IV fentanyl for peri-procedural analgesia
  Interventions: Drug: Fentanyl; Drug: Lidocaine; Drug: Midazolam

INTERVENTIONS:
Other: Removal of Fentanyl from peri-procedural analgesia — Removal of Fentanyl from peri-procedural analgesia (which is otherwise routinely given for PCI)
  Arms: PCI without IV opiate
Drug: Fentanyl — IV peri-procedural analgesia
  Arms: PCI with IV opiate
Drug: Lidocaine — Local Anesthetic
Drug: Midazolam — IV sedation

SUMMARY:
With potent analgesic properties, perceived hemodynamic benefits and limited alternatives, opiates are the analgesic mainstay for acute coronary syndrome (ACS) patients reporting peri-procedural pain or nitrate-resistant chest pain. However, large observational studies suggest that opiate administration during ACS may result in adverse cardiovascular outcomes. Complimenting this, a number of recent mechanistic studies have demonstrated delayed and attenuated effects of oral dual anti-platelet therapy (DAPT) on platelet inhibition endpoints among subjects receiving intravenous morphine. These studies support the hypothesis that morphine delays the gastrointestinal absorption of DAPT medications. However, no data exist on the impact of intravenous fentanyl, a systemic opioid analgesic routinely administered during percutaneous coronary intervention (PCI) procedures, on the platelet inhibition effects of DAPT. The investigators hypothesize that, similar to morphine, fentanyl administered at the time of PCI will reduce and delay the effect of DAPT on platelet function. As such, the primary aim of this study is to test the impact of intravenous fentanyl on residual platelet reactivity by randomizing patients undergoing PCI to a strategy of peri-procedural benzodiazepine plus non-systemic local analgesia or to the current standard of benzodiazepine plus intravenous fentanyl. Given the critical need for rapid and robust inhibition of platelet function during PCI, this trial has true potential to change clinical practice, particularly if the investigators demonstrate reduced DAPT absorption and elevated residual platelet reactivity among patients receiving fentanyl during PCI.

ELIGIBILITY:
Inclusion Criteria:

* undergoing clinically indicated PCI; >18 years of age; able for PO medications and to provide informed consent

Exclusion Criteria:

* pregnant; any DAPT(clopidogrel, prasugrel, ticagrelor) within 14 days of enrollment; known coagulation disorders; active treatment with oral anticoagulant or low molecular weight heparin; impaired renal or hepatic function; platelets < 100 x10 3 /mcl; planned use of Glycoprotein 2b3a for PCI; Prior Trans Arterial Valve Replacement (TAVR) or planned TAVR post PCI; and contraindications to ticagrelor or opiates.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W McEvoy, MBBCh MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital and University School of Medicicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ibrahim K, Shah R, Goli RR, Kickler TS, Clarke WA, Hasan RK, Blumenthal RS, Thiemann DR, Resar JR, Schulman SP, McEvoy JW. Fentanyl Delays the Platelet Inhibition Effects of Oral Ticagrelor: Full Report of the PACIFY Randomized Clinical Trial. Thromb Haemost. 2018 Aug;118(8):1409-1418. doi: 10.1055/s-0038-1666862. Epub 2018 Jul 4. PMID 29972861
- [Derived] Ibrahim K, Goli RR, Shah R, Resar JR, Schulman SP, McEvoy JW. Effect of intravenous fentanyl on ticagrelor absorption and platelet inhibition among patients undergoing percutaneous coronary intervention: Design, rationale, and sample characteristics of the PACIFY randomized trial. Contemp Clin Trials. 2018 Jan;64:8-12. doi: 10.1016/j.cct.2017.11.011. Epub 2017 Nov 21. PMID 29170073
- [Derived] McEvoy JW, Ibrahim K, Kickler TS, Clarke WA, Hasan RK, Czarny MJ, Keramati AR, Goli RR, Gratton TP, Brinker JA, Chacko M, Hwang CW, Johnston PV, Miller JM, Trost JC, Herzog WR, Blumenthal RS, Thiemann DR, Resar JR, Schulman SP. Effect of Intravenous Fentanyl on Ticagrelor Absorption and Platelet Inhibition Among Patients Undergoing Percutaneous Coronary Intervention: The PACIFY Randomized Clinical Trial (Platelet Aggregation With Ticagrelor Inhibition and Fentanyl). Circulation. 2018 Jan 16;137(3):307-309. doi: 10.1161/CIRCULATIONAHA.117.031678. Epub 2017 Oct 18. No abstract available. PMID 29046319

RESULTS

PARTICIPANT FLOW:
Groups:
- PCI Without Intranvenous (IV) Opiate: IV midazolam and Local Anesthetic, with removal of IV fentanyl from peri-procedural analgesia (which is otherwise routinely given)
  Removal of Fentanyl from peri-procedural analgesia: Removal of Fentanyl from peri-procedural analgesia (which is otherwise routinely given for percutaneous coronary intervention [PCI])
  Lidocaine: Local Anesthetic
  Midazolam: IV sedation
Period: Overall Study
Arm/Group | PCI Without Intranvenous (IV) Opiate | PCI With IV Opiate
Started | 105 | 107
Completed | 105 | 107
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCI Without IV Opiate | PCI With IV Opiate | Total
Number analyzed (Participants) | 105 | 107 | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9.3) | 63 (10.2) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 25 | 67
  Male | 63 | 82 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 15 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 17 | 36
  White | 79 | 75 | 154
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 105 | 107 | 212
Platelet count [Mean (Standard Deviation); unit: K/cu mm] | 230 (59) | 223 (71) | 226 (65)

OUTCOME MEASURES:

1. Primary Outcome: Ticagrelor Pharmacokinetics
Description: Area under the curve for Ticagrelor Absorption
Time Frame: Measured over 24 hours (at 0, 0.5, 1, 2, 4, and 24 hours)
Population: Only the subgroup (n=70) of enrolled participants who required PCI and were loaded with ticagrelor had information on the primary endpoint
Measure: Mean (Standard Error); unit: ng*hr/mL
Arm/Group | PCI Without IV Opiate | PCI With IV Opiate
Number analyzed (Participants) | 35 | 35
ng*hr/mL | 3301 (271) | 2107 (301)

2. Secondary Outcome: Single Time-point Platelet Reactivity Using Verify Now
Description: Blood test of Platelet Cell Reactivity using Verify Now (P2Y12 Reactivity Units)
Time Frame: Measured at 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: PRUs
Arm/Group | PCI Without IV Opiate | PCI With IV Opiate
Number analyzed (Participants) | 35 | 35
PRUs | 78 (72) | 112 (95)

3. Secondary Outcome: Platelet Reactivity Using Light Transmission Aggregometry
Description: Blood test of Platelet Cell Reactivity using Light Transmission Aggregometry (reported as percent of baseline aggregation in response to adenosine diphosphate stimulation)
Time Frame: Measured at 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of baseline aggregation
Arm/Group | PCI Without IV Opiate | PCI With IV Opiate
Number analyzed (Participants) | 35 | 35
percentage of baseline aggregation | 27.5 (14.4) | 39.3 (8.7)

4. Secondary Outcome: Patient Self-reported Pain
Description: Patient self report of pain using a visual analog scale (VAS). Scale ranges from 0 to 10 with 0 being "No pain" and 10 being "Most severe pain".
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PCI Without IV Opiate | PCI With IV Opiate
Number analyzed (Participants) | 105 | 107
units on a scale | 2.3 (3.1) | 1.5 (2.3)

ADVERSE EVENTS:
Time Frame: Adverse event data (specifically pain and anxiety reports from participants) were collected on the day of the procedure during which each participant was under study.
Arm/Group | PCI Without IV Opiate | PCI With IV Opiate
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/107
Serious Adverse Events (participants affected / at risk) | 13/105 | 7/107
Other Adverse Events (participants affected / at risk) | 0/105 | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCI Without IV Opiate (N=105) | PCI With IV Opiate (N=107)
Pain >5/10 (General disorders) | 13 (13) | 7 (7)

LIMITATIONS AND CAVEATS:
Small sample, surrogate endpoints

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT02683707/Prot_SAP_000.pdf